CLINICAL TRIAL: NCT00086463
Title: A Safety and Pilot Efficacy Trial of Iloprost Inhaled Solution as Add-On Therapy With Bosentan in Subjects With PAH
Brief Title: Trial of Iloprost Inhaled Solution as Add-On Therapy With Bosentan in Subjects With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STEP STUDY; STEP; Pulmonary Hypertension; Pulmonary Artery; Cotherix
Record Dates: First submitted 2004-07-01; First posted 2004-07-05 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Pulmonary Arterial Hypertension; Ayerza Syndrome; Pulmonary Hypertension
Keywords: STEP; PAH; iloprost; inhalation; prostacyclin
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Respiratory Aspiration | interventions — Iloprost

INTERVENTIONS:
Drug: Iloprost or placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Iloprost in subjects that have Pulmonary Arterial Hypertension who are concurrently taking bosentan (Tracleer TM).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled study in subjects with Pulmonary Arterial Hypertension (PAH) with an NYHA Class of III or IV who are receiving conventional therapy and bosentan. Subjects who fulfill the inclusion and exclusion criteria will be randomized to study drug (active or placebo) at a frequency of 6-9 inhalations per day for 12 weeks and will continue conventional therapy and bosentan. At the end of the double-blind phase study, open label Iloprost will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAH due to PPH, connective tissue disease, HIV, or repaired (≥ 1 year) ASD, VSD, or PDA
* NYHA Functional Class III or IV
* On bosentan for at least 16 weeks, with the dose stable (maximum dose 125 mg BID) for at least 8 weeks
* Age 12-75 years, of either gender
* Six minute walk distance 100-425 meters at Baseline

Exclusion Criteria:

* Any new long-term treatment for PAH added within the last 4 weeks
* Any therapy with a PDE (phosphodiesterase), L -arginine or a prostaglandin, concurrently, or within the last 4 weeks
* PAH related to chronic thromboembolic disease, portopulmonary disease, or any etiology other than PPH, connective tissue disease, HIV, or repaired ASD, VSD, or PDA

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hsu, M.D., Study Director — CoTherix
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Medical Center, La Jolla, California
  - Stanford University Medical Center, Palo Alto, California
  - UCSF Medical Center, San Francisco, California
  - Harbor-UCLA Medical Center, Torrance, California
  - The Children's Hospital, Denver, Colorado
  - University of Colorado HSC, Denver, Colorado
  - Rush Heart Institute, Center for Pulmonary Heart Disease, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Latter Day Saints Hospital, Salt Lake City, Utah

REFERENCES:
- [Background] Olschewski H, Simonneau G, Galie N, Higenbottam T, Naeije R, Rubin LJ, Nikkho S, Speich R, Hoeper MM, Behr J, Winkler J, Sitbon O, Popov W, Ghofrani HA, Manes A, Kiely DG, Ewert R, Meyer A, Corris PA, Delcroix M, Gomez-Sanchez M, Siedentop H, Seeger W; Aerosolized Iloprost Randomized Study Group. Inhaled iloprost for severe pulmonary hypertension. N Engl J Med. 2002 Aug 1;347(5):322-9. doi: 10.1056/NEJMoa020204. PMID 12151469